CLINICAL TRIAL: NCT02789787
Title: Clinical Effectiveness of Late Maxillary Protraction for Cleft Lip and Palate
Acronym: PROTRACTSURG
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Seattle Children's Hospital (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Stephen Yen, Associate Professor, University of Southern California
Other Study IDs: 5U01DE022937-04 (NIH)
Record Dates: First submitted 2016-05-09; First posted 2016-06-03 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Cleft Lip and Palate
Keywords: Cleft Lip; Palate; Class III; Malocclusion; Protraction
MeSH Terms: conditions — Cleft Lip; Malocclusion | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Maxillary protraction: Early adolescents (11 - 14 yrs) with cleft lip and palate and Cl III malocclusion
  Interventions: Procedure: Maxillary Protraction
- Orthognathic surgery: Late adolescents to young adults (16-21 years) with cleft lip and palate and Cl III malocclusion
  Interventions: Procedure: Orthognathic Surgery

INTERVENTIONS:
Procedure: Maxillary Protraction — "Maxillary protraction" is an alternative non-surgical approach to correct the Cl III malocclusion. At ages 11- 14, the maxillary sutures have not fused and can be mobilized by alternating weekly expansion and constriction with a rapid palatal expander (RPE), thereby allowing the maxilla to be protracted in order to correct the underbite. This treatment is offered to the patients, age 11-14, who have the Cl III malocclusion with or without cleft lip and palate.
  Groups: Maxillary protraction
Procedure: Orthognathic Surgery — The orthognathic surgery is the current standard of care for treating the Cl III malocclusion after pubertal growth. This treatment is offered to the patients, after pubertal growth, who have the Cl III malocclusion with or without cleft lip and palate.
  Other Names: LeFort 1 maxillary advancement surgery
  Groups: Orthognathic surgery

SUMMARY:
Patients with cleft lip and palate frequently develop Class III (Cl III) malocclusions or underbites following early cleft repair surgeries. This clinical trial compares the current standard of care for treating the Cl III malocclusion, orthognathic (jaw) surgery after pubertal growth (16-21 years), with an alternative orthopedic approach to protract the maxilla during adolescence (11-14 years). At Children's Hospital Los Angeles(CHLA), early adolescents with cleft lip and palate and Cl III malocclusion are offered an alternative non-surgical approach to correct the malocclusion called "maxillary protraction". Prior to age 14, the maxillary sutures have not fused and can be mobilized by alternating weekly expansion and constriction with a rapid palatal expander (RPE), thereby allowing the upper jaw (maxilla) to be pulled forward (protracted) to correct the underbite. This prospective parallel cohort study will assess the patients undergoing treatment for the Cl III malocclusion by either orthognathic surgery or maxillary protraction at four data collection time points during treatment. The data includes digitized study models, photographs and radiographs, quality of life surveys (SF12, YQOL), parent surveys (ASEBA), treatment cost, periodontal measurements and treatment complications. The study design is a descriptive cohort study that examines the success of treatment (% not requiring a second surgery), the dental and skeletal changes associated with treatment, the stability of treatment and the behavioural/adaptive factors (ASEBA) that contribute to success and lack of success for each treatment. The primary trial will be conducted at Children's Hospital Los Angeles and a pilot study to confirm translation to different settings will be conducted at Seattle Children's Hospital.

DETAILED DESCRIPTION:
Rationale: Cleft lip and palate is the most common facial birth defect. Patients with cleft lip and palate frequently develop Class III (Cl III) malocclusion or underbites for which the current standard of care to treat the Cl III malocclusion is orthognathic (jaw) surgery. Orthognathic surgery is performed late in a teenager's life after pubertal growth is complete, has a long recovery period, has risks for segment loss and nerve injury and is expensive to the insurers. Moreover, the surgical correction can relapse and require a second jaw surgery.

Intervention: The current standard of care for correcting a Cl III malocclusion is orthognathic surgery after pubertal growth is complete. At Children's Hospital, early adolescents (11 - 14 yrs) with cleft lip and palate and Cl III malocclusion are offered an alternative non-surgical approach to correct the malocclusion called "maxillary protraction". At ages 11- 14, the maxillary sutures have not fused and can be mobilized by alternating weekly expansion and constriction with a rapid palatal expander (RPE), thereby allowing the upper jaw (maxilla) to be pulled forward (protracted) in order to correct the underbite.

Purpose: This study will compare the occlusal, photographic, radiographic, periodontal and quality of life data collected at four different timepoints from patients who were treated for the correction of their Cl III malocclusion by either LeFort I maxillary advancement surgery or non-surgical maxillary protraction.

Study Population: The inclusion criteria are patients who are diagnosed with isolated cleft lip and palate with Cl III malocclusion and who, at the time of enrollment, do not have any medical condition which will prevent them from undergoing orthognathic surgery or maxillary protraction procedures. The two study groups differ in age and treatment. One group of patients, ages 11 -14 years of age, chose to undergo maxillary protraction via sutural loosening for correction of Cl III malocclusion. The other group of patients, ages 16 and 21 years, elected to undergo orthognathic surgery for correction of Cl III malocclusion.

Study Methodology: This is a non-randomized prospective parallel cohort study that follows the treatment outcomes of approximately 100 patients with cleft lip and palate and Cl III malocclusion who are treated with maxillary protraction at about a maximal age of 14 years (target N=50) vs. orthognathic surgery at a maximal age of 21 years (target N=50).

Description of Treatment Arms: The first treatment arm consists of participants who have chosen to undergo the orthodontic (non-surgical) maxillary protraction procedure. The second treatment arm consists of participants who have chosen to undergo the orthognathic (jaw) surgical procedure.

Outcomes: The outcomes measured in both groups will be bite correction (GOSLON yardstick), facial esthetics, changes in cephalometric x-ray measurements, youth quality of life (YQOL), psychological/behavioral assessment surveys (ASEBA), cost, periodontal health, complications and stability of treatment.

Follow-up: Participants in both arms of the study (protraction vs. surgery) will have data collected prior to, during, immediately after, and 1 year after treatment.

Statistics and Plans for Analysis: The % of patients requiring further surgery and the reasons for the relapse or incomplete treatment will be examined using the collected data. The investigators will examine factors that are associated with the successful outcomes for each treatment and adjust for these factors in the models.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonsyndromic cleft lip and palate and Class III malocclusion
* Age 11-14 for maxillary protraction, Age 16-21 for LeFort I single jaw surgery.

Exclusion Criteria:

* Cognitive delay;
* Mandibular asymmetry;
* Mandibular prognathism;
* 2-jaw cants;
* Non-grafted alveolar cleft;
* Inability or unwillingness to have clinical radiographs, photographs, or dental impressions taken;
* History of therapeeutic radiation treatment to the mazilla or mandible;
* Pregnancy; if participants become pregnant during the study they will be withdrawn.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with nonsyndromic cleft lip and palate who have a Cl III malocclusion
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Bite correction of digitized models. | Approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The metric for comparing the difference in bite using study models from patients with cleft lip and palate is the "GOSLON Yardstick" which can rate antero-posterior as well as transverse positions.

SECONDARY OUTCOMES:
Cephalometric radiographs | The four timepoints during approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The cephalometric radiographs from the different time points are stored in Dolphin imaging software and digitized for orthodontic and surgical cephalometric analyses. This type of analysis can examine differences between skeletal vs. dental changes between time points.
Facial attractive rating of photographs | The four timepoints during approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The pre-treatment and post-treatment facial photographs of all of the patients in the study will be randomly presented for rating using an analog scale for facial attractiveness. The photographs are presented in a secure database file within the hospital to lay and clinician raters for evaluating the photographs. This type of rating survey can provide data on amount and direction of facial change with each treatment.
Costs of treatments | At the end of approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The number of visits and current procedural terminology(CPT) codes for the visits will be used to define cost units. The actual costs for CHLA and SCH will be calculated by assigning the hospital charges for those CPT codes.
12-Item Short Form Health Survey (SF-12) developed by the Rand Corporation | The four timepoints during approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The SF-12 is a short form standardized instrument for medical outcome study.
Youth Quality of Life (YQOL) survey designed by the Seattle Quality of Life Group | The four timepoints during approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The YQOL instrument assesses multidimensionally the generic quality of life of youth ages 11-18 years of age. YQOL includes both generic and condition-specific measures.
Achenbach System of Empirically Based Assessment (ASEBA) | The four timepoints during approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The ASEBA offers a comprehensive approach to assessing adaptive and maladaptive functioning.These surveys are given to the parents of the patients in the study in order to provide a behavioural assessment of their child.
Periodontal measurements | Approximately 36-48 months for maxillary protraction patients and approximately 36-42 months for patients undergoing orthognathic surgery.
  The periodontal condition of the premolars and molars normally used for maxillary protraction are evaluated using bleeding index, plaque scores, probe depth and mobility scores.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Yen, DMD, PhD, Principal Investigator — CHLA; Jane Atkinson, Study Director — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All of the participant data collected during the trial after deidentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Chung EH, Borzabadi-Farahani A, Yen SL. Clinicians and laypeople assessment of facial attractiveness in patients with cleft lip and palate treated with LeFort I surgery or late maxillary protraction. Int J Pediatr Otorhinolaryngol. 2013 Sep;77(9):1446-50. doi: 10.1016/j.ijporl.2013.05.042. Epub 2013 Jul 18. PMID 23871270
- [Background] Yen SL. Protocols for Late Maxillary Protraction in Cleft Lip and Palate Patients at Childrens Hospital Los Angeles. Semin Orthod. 2011 Jun 1;17(2):138-148. doi: 10.1053/j.sodo.2011.01.001. PMID 21765629
- [Background] McIlvaine E, Borzabadi-Farahani A, Lane CJ, Azen SP, Yen SL. Apriori feasibility testing of randomized clinical trial design in patients with cleft deformities and Class III malocclusion. Int J Pediatr Otorhinolaryngol. 2014 May;78(5):725-30. doi: 10.1016/j.ijporl.2014.01.006. Epub 2014 Feb 12. PMID 24630053
- [Result] Borzabadi-Farahani A, Lane CJ, Yen SL. Late maxillary protraction in patients with unilateral cleft lip and palate: a retrospective study. Cleft Palate Craniofac J. 2014 Jan;51(1):e1-e10. doi: 10.1597/12-099. Epub 2012 Dec 13. PMID 23237432